CLINICAL TRIAL: NCT00464399
Title: A Pilot Study to Evaluate Feasibility and Safety of Early Switch to Everolimus From Cyclosporine in de Novo Renal Transplant
Brief Title: Feasibility and Safety of Early Switch to Everolimus From Cyclosporine in de Novo Renal Transplant Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ANO01
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: De Novo Renal Transplantation
Keywords: De novo renal transplantation; CNI-free protocol; adults; everolimus; rejections
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: everolimus

SUMMARY:
To evaluate the safety and tolerability of early switch to everolimus from cyclosporine A in de novo renal transplant recipients by assessing rejection rate everolimus trough levels, other safety laboratory variables and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged above 18 years.
* Patients having received their first or second single renal transplant from deceased or living donor
* Patient willing and capable of giving written informed consent for study participation
* Patients treated with as induction therapy at the time of transplantation
* Patients maintained on a triple immunosuppressive regime consisting of cyclosporine (C-0 h between 100-250 ng/ml or a C-2 h between 900-1100 ng/ml), Enteric coated mycophenolate sodium (EC-MPS), minimum dose 1080 mg and corticosteroids, minimum dose 10 mg
* Patients without any biopsy proven acute rejection episode or treatment for any acute rejection since the transplant
* Females capable of becoming pregnant must have a negative pregnancy test prior to the switch to everolimus and are required to practice a medically approved method of birth control for the duration of the study and a period of 8 weeks following discontinuation of study medication, even where there has been a history of infertility.

Exclusion Criteria:

* Recipient of multi-organ transplants, and or previously transplanted with any other organ different from a kidney transplant
* Patients with antibodies towards the donor kidney above 30%
* Patients receiving a renal transplant from HLA-identical sibling
* Presence of hyper sensitivity to drugs similar to everolimus ( e.g. macrolides)
* Patient with past (within the last two years) or present malignancy other than excised basal cell or squamous cell carcinoma of the skin
* Patients who are recipients of AB0 incompatible transplants
* Patients with unsuitable laboratory values
* Patients with ongoing wound healing problems or other severe surgical complication in the opinion of the investigator
* Patient with a current severe major local or systemic infection
* Patients requiring dialysis and/or having a calculated glomerular filtration rate (Cockcroft-Gault) < 20 ml/min
* Presence of intractable immunosuppressant complications or side effects (e.g., severe gastrointestinal adverse events) at the time of the switch
* Patients who are HIV positive or Hepatitis B surface antigen positive or Hepatitis C virus positive. Recipients of organs from donors who test positive for Hepatitis B surface antigen or Hepatitis C are excluded.
* Evidence of severe liver disease

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-09; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Biopsy proven acute rejections or treatment for acute rejections from the time of the conversion from cyclosporine based regimen to a cyclosporine free treatment with everolimus 7 weeks ± 7 days after transplantation until completion of 7 weeks after

SECONDARY OUTCOMES:
Efficacy assessed by graft and patients survival from the time of conversion 7 weeks ± 7 days until the end of follow-up 12 months after transplantation
Pharmacokinetics assessed by blood samples for everolimus concentration , cyclosporine concentrations
Safety assessed by blood sampling for Hemoglobin, white blood cells (WBC), platelets, s-creatinine, ASAT, ALAT, ALP bilirubin, S-Na, S-K, S-Ca, S-P. S-Urea, S-creatin phosphokinase (S-CPK), u-alb/creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site,, Oslo, Norway

REFERENCES:
- [Result] Holdaas H, Bentdal O, Pfeffer P, Mjornstedt L, Solbu D, Midtvedt K. Early, abrupt conversion of de novo renal transplant patients from cyclosporine to everolimus: results of a pilot study. Clin Transplant. 2008 May-Jun;22(3):366-71. doi: 10.1111/j.1399-0012.2008.00795.x. Epub 2008 Feb 12. PMID 18279419